CLINICAL TRIAL: NCT03776669
Title: Laparoscopic Sleeve Gastrectomy With or Without Hiatal Hernia Repair in Morbidly Obese Patients: a Single-center Randomized Controlled Trial
Brief Title: Laparoscopic Sleeve Gastrectomy With or Without Hiatal Hernia Repair in Morbidly Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201810017RINB
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Morbid Obesity; Hiatal Hernia; Gastroesophageal Reflux Disease; Sleeve Gastrectomy
Keywords: Morbid obesity; Hiatal hernia; Gastroesophageal reflux disease; High resolution impedance manometry
MeSH Terms: conditions — Obesity, Morbid; Hernia, Hiatal; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSG alone (Active Comparator): Intervention: laparoscopic sleeve gastrectomy alone.
  LSG will be performed laparoscopically via a 5-port technique. The greater omentum is dissected by using the 5-mm laparoscopic LigaSure or Harmonic from 4 cm proximal to the pyloric ring to the angle of His. Sleeve calibration is done by a 36-French bougie inserted along the lesser curvature. Then the stomach is transected with sequential firings of linear green, gold, and blue 60 mm staplers starting about 4 cm proximal to the pylorus and ending approximately 2 cm distal to the left of the esophagus. The staple-line of the remnant gastric tube is oversewn with 3-0 V-Loc to prevent leakage and hemorrhage.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy alone
- LSG + HHR (Experimental): Intervention: concomitant laparoscopic sleeve gastrectomy + hiatal hernia repair.
  The surgical detail of LSG is the same as described in "LSG alone" arm, and the surgical detail of HHR is described as below.
  The hiatus is approached from the right side of the EGJ, through the lesser omentum. The hiatal defect is repaired by 1-0 Surgilon interruptedly, and then a commercialized "U-shaped" Biodesign Hiatal Hernia Graft is placed to the EGJ to cover the posterior side but spare the anterior side of the hiatus. Care must be taken to avoid direct contact of mesh to the esophagus to avoid any unnecessary complication. After the mesh is appropriately placed and oriented, 2 ml of TISSEEL solution for sealant is applied all over the mesh for fixation.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy + Hiatal hernia repair

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy + Hiatal hernia repair — To evaluate the role of concomitant hiatal hernia repair in laparoscopic sleeve gastrectomy for morbidly obese patients.
  Arms: LSG + HHR
Procedure: Laparoscopic sleeve gastrectomy alone — Current mainstay and standard surgical treatment for morbidly obese patients.
  Arms: LSG alone

SUMMARY:
Background:

Obesity and hiatal hernia are both risk factors of gastroesophageal reflux disease (GERD), and the incidence of hiatal hernia is much higher in morbidly obese patients. Many believe that higher intra-abdominal pressure with higher esophagogastric junction (EGJ) pressure gradient in morbidly obese patients is the main mechanism accounting for the occurrence of GERD. Hiatal hernia, on the other hand, is associated with structure abnormality of EGJ. Sleeve gastrectomy (SG) has been becoming a standalone bariatric surgery for decades, and it has been proved to effectively induce long-term weight loss in morbidly obese patients. Some studies found morbidly obese patients benefited from resolution of GERD after SG, however, other studies had the opposite findings. Some morbidly obese patients had aggravating GERD or de novo GERD after SG. The mechanism is still unclear now. It might result from removal of fundus and sling muscular fibers of EGJ, increased intra-gastric pressure (IIGP), and hiatal hernia after surgery. High resolution impedance manometry (HRIM) is used to access esophageal and EGJ function objectively. Impedance reflux was more frequently observed in patients having gastroesophageal reflux (GER) symptoms after SG. In addition, previous studies also found decreased EGJ resting pressure, decreased length of lower esophageal sphincter (LES), and presence of hiatal hernia were associated with more GERD after SG.

Objective:

To evaluate the long-term EGJ function and GERD in morbidly obese patients with hiatal hernia receiving laparoscopic sleeve gastrectomy (LSG) with or without hiatal hernia repair (HHR).

DETAILED DESCRIPTION:
Patients and methods:

A total of 70 patients will be recruited and randomized to two groups with a 1:1 allocation ratio. Patients in the control group receive LSG alone and in the experimental group receive LSG with HHR. All subjects should provide basic clinical and demographic information, be evaluated for GER symptoms using GerdQ score, sign informed consent, and complete preoperative abdominal computed tomography (CT) scan, esophagogastroduodenoscopy (EGD), and HRIM. Outpatient follow-up would be arranged 1 weeks after discharge, then 1 month, 3 months, 6 months, and 12 months after surgery. Weight change and GER symptoms will be evaluated at every outpatient visit. Abdominal CT scan, EGD, and HRIM will be performed 12 months after surgery.

Expected results:

Less reflux esophagitis, less impedance reflux episodes, lower incidence of hiatal hernia, higher EGJ resting pressure, and longer LES length should be observed in morbidly obese patients receiving LSG with HHR at 12-month follow-up, using EGD and HRIM as evaluation tools. Furthermore, lower GerdQ score should be observed in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with:

  1. Body mass index (BMI) ≧ 35, or
  2. 30 ≦ BMI < 35, with inadequately controlled type 2 diabetes mellitus (T2DM) or metabolic syndrome, or
  3. T2DM with BMI ≧ 32.5, or
  4. T2DM with BMI between 27.5 and 32.5 not well controlled by medication, especially for those with major cardiovascular risk.
* Age: 20 to 65 years old.
* Hiatal hernia diagnosed by either:

  1. HRIM: defined as the distance between low esophageal sphincter (LES) and crural diaphragm (CD) equal to or greater than 2 cm. (LES-CD ≧ 2 cm)
  2. EGD: defined as the apparent separation between the squamocolumnar junction and the diaphragmatic impression is greater than 2 cm.

Exclusion Criteria:

* Prior major gastrointestinal (GI) tract surgery.
* Bleeding tendency.
* American Society of Anesthesiologists physical status (ASA) ≧ class III.
* Pregnancy or lactating women.
* Allergy to contrast medium for CT scan.
* Concomitantly untreated or uncontrolled endocrine disease.
* Alcohol or drug abuse.
* Mental, behavioral, and neurodevelopmental disorders.

  1. Patients who possess "National Health Insurance (NHI) Major Illness/Injury Certificate" for ICD-10-CM codes F01-F99. (ICD: International Classification of Diseases; CM: Clinical Modification)
  2. Patients who have been hospitalized in psychiatric ward in the recent one year.
* Type IV hiatal hernia.
* Moderate to severe reflux esophagitis (LA classification grade B/C/D) refractory to medical treatment.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-01-09 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-12-17 (Estimated)

PRIMARY OUTCOMES:
De novo reflux esophagitis | Within 12 months after surgery if symptomatic or at 12 months if asymptomatic.
  Los angles classification grade B/C/D reflux esophagitis diagnosed by esophagogastroduodenoscopy.

SECONDARY OUTCOMES:
Impedance reflux | 12 months after the surgery
  Impedance reflux after single swallow by high resolution impedance manometry
Esophagogastric junction (EGJ) resting pressure | 12 months after the surgery
  Measured by high resolution impedance manometry
Lower esophageal sphincter (LES) length | 12 months after the surgery
  Measured by high resolution impedance manometry
De novo or aggravating hiatal hernia | 12 months after the surgery (or within 12 months after surgery if symptomatic )
  Diagnosed by high resolution impedance manometry or esophagogastroduodenoscopy.
GerdQ score | At 1 week (± 1 week) after discharge, then 1 month (± 2 weeks), 3 months (± 1 month), 6 months (± 1 month), and 12 months (± 1 month) after surgery.
  Questionnaire for gastroesophageal reflux symptoms
Post-operative complication | Within 30 days of surgery
  Defined as complication ≧ grade III Clavien-Dindo classification
Mesh-related complication | Within 12 months after surgery
  infection, allergic reaction, intestinal complication, fistula formation, seroma formation, hematoma, recurrence of tissue defect, dysphagia, esophageal erosion or perforation.

CONTACTS AND LOCATIONS:
Overall Officials: PoChu Lee, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no individual patient data (IPD) sharing plan now.

REFERENCES:
- [Background] Che F, Nguyen B, Cohen A, Nguyen NT. Prevalence of hiatal hernia in the morbidly obese. Surg Obes Relat Dis. 2013 Nov-Dec;9(6):920-4. doi: 10.1016/j.soard.2013.03.013. Epub 2013 Apr 19. PMID 23810611
- [Background] Santonicola A, Angrisani L, Cutolo P, Formisano G, Iovino P. The effect of laparoscopic sleeve gastrectomy with or without hiatal hernia repair on gastroesophageal reflux disease in obese patients. Surg Obes Relat Dis. 2014 Mar-Apr;10(2):250-5. doi: 10.1016/j.soard.2013.09.006. Epub 2013 Sep 20. PMID 24355324
- [Background] Soricelli E, Iossa A, Casella G, Abbatini F, Cali B, Basso N. Sleeve gastrectomy and crural repair in obese patients with gastroesophageal reflux disease and/or hiatal hernia. Surg Obes Relat Dis. 2013 May-Jun;9(3):356-61. doi: 10.1016/j.soard.2012.06.003. Epub 2012 Jun 19. PMID 22867558
- [Background] Mahawar KK, Carr WR, Jennings N, Balupuri S, Small PK. Simultaneous sleeve gastrectomy and hiatus hernia repair: a systematic review. Obes Surg. 2015 Jan;25(1):159-66. doi: 10.1007/s11695-014-1470-0. PMID 25348434
- [Background] Crawford C, Gibbens K, Lomelin D, Krause C, Simorov A, Oleynikov D. Sleeve gastrectomy and anti-reflux procedures. Surg Endosc. 2017 Mar;31(3):1012-1021. doi: 10.1007/s00464-016-5092-6. Epub 2016 Jul 20. PMID 27440196
- [Background] Braghetto I, Lanzarini E, Korn O, Valladares H, Molina JC, Henriquez A. Manometric changes of the lower esophageal sphincter after sleeve gastrectomy in obese patients. Obes Surg. 2010 Mar;20(3):357-62. doi: 10.1007/s11695-009-0040-3. Epub 2009 Dec 15. PMID 20013071
- [Background] DuPree CE, Blair K, Steele SR, Martin MJ. Laparoscopic sleeve gastrectomy in patients with preexisting gastroesophageal reflux disease : a national analysis. JAMA Surg. 2014 Apr;149(4):328-34. doi: 10.1001/jamasurg.2013.4323. PMID 24500799
- [Background] Oor JE, Roks DJ, Unlu C, Hazebroek EJ. Laparoscopic sleeve gastrectomy and gastroesophageal reflux disease: a systematic review and meta-analysis. Am J Surg. 2016 Jan;211(1):250-67. doi: 10.1016/j.amjsurg.2015.05.031. Epub 2015 Aug 14. PMID 26341463
- [Background] Soricelli E, Casella G, Rizzello M, Cali B, Alessandri G, Basso N. Initial experience with laparoscopic crural closure in the management of hiatal hernia in obese patients undergoing sleeve gastrectomy. Obes Surg. 2010 Aug;20(8):1149-53. doi: 10.1007/s11695-009-0056-8. Epub 2010 Jan 5. PMID 20049652
- [Background] Ruscio S, Abdelgawad M, Badiali D, Iorio O, Rizzello M, Cavallaro G, Severi C, Silecchia G. Simple versus reinforced cruroplasty in patients submitted to concomitant laparoscopic sleeve gastrectomy: prospective evaluation in a bariatric center of excellence. Surg Endosc. 2016 Jun;30(6):2374-81. doi: 10.1007/s00464-015-4487-0. Epub 2015 Oct 1. PMID 26428202
- [Background] Samakar K, McKenzie TJ, Tavakkoli A, Vernon AH, Robinson MK, Shikora SA. The Effect of Laparoscopic Sleeve Gastrectomy with Concomitant Hiatal Hernia Repair on Gastroesophageal Reflux Disease in the Morbidly Obese. Obes Surg. 2016 Jan;26(1):61-6. doi: 10.1007/s11695-015-1737-0. PMID 25990380
- [Background] Tutuian R, Vela MF, Shay SS, Castell DO. Multichannel intraluminal impedance in esophageal function testing and gastroesophageal reflux monitoring. J Clin Gastroenterol. 2003 Sep;37(3):206-15. doi: 10.1097/00004836-200309000-00004. PMID 12960718
- [Background] Kahrilas PJ, Bredenoord AJ, Fox M, Gyawali CP, Roman S, Smout AJ, Pandolfino JE; International High Resolution Manometry Working Group. The Chicago Classification of esophageal motility disorders, v3.0. Neurogastroenterol Motil. 2015 Feb;27(2):160-74. doi: 10.1111/nmo.12477. Epub 2014 Dec 3. PMID 25469569
- [Background] Suter M, Dorta G, Giusti V, Calmes JM. Gastro-esophageal reflux and esophageal motility disorders in morbidly obese patients. Obes Surg. 2004 Aug;14(7):959-66. doi: 10.1381/0960892041719581. PMID 15329186
- [Background] Mion F, Tolone S, Garros A, Savarino E, Pelascini E, Robert M, Poncet G, Valette PJ, Marjoux S, Docimo L, Roman S. High-resolution Impedance Manometry after Sleeve Gastrectomy: Increased Intragastric Pressure and Reflux are Frequent Events. Obes Surg. 2016 Oct;26(10):2449-56. doi: 10.1007/s11695-016-2127-y. PMID 26956879
- [Background] Jones R, Junghard O, Dent J, Vakil N, Halling K, Wernersson B, Lind T. Development of the GerdQ, a tool for the diagnosis and management of gastro-oesophageal reflux disease in primary care. Aliment Pharmacol Ther. 2009 Nov 15;30(10):1030-8. doi: 10.1111/j.1365-2036.2009.04142.x. Epub 2009 Sep 8. PMID 19737151
- [Background] Bredenoord AJ, Fox M, Kahrilas PJ, Pandolfino JE, Schwizer W, Smout AJ; International High Resolution Manometry Working Group. Chicago classification criteria of esophageal motility disorders defined in high resolution esophageal pressure topography. Neurogastroenterol Motil. 2012 Mar;24 Suppl 1(Suppl 1):57-65. doi: 10.1111/j.1365-2982.2011.01834.x. PMID 22248109